CLINICAL TRIAL: NCT03364621
Title: Comprehensive Genomic Profiling of Colorectal Cancer Patients With Isolated Liver Metastases to Understand Response & Resistance to Cancer Therapy
Acronym: COMPARISON
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Terry Fox Research Institute (Other); British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: COMPARISON-001
Record Dates: First submitted 2017-11-09; First posted 2017-12-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; Colorectal Cancer Metastatic; Hepatic Metastases
Keywords: Liver resection; Metastasis; Molecular profiling; Epigenetic analysis; Genomic analysis; Sequencing
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival primary tumor tissue, fresh liver tumor tissue, baseline tube whole blood, serial 4x tube of whole blood every 3-6 months until disease relapse or 2 years post-liver resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Metastatic Colorectal Cancer with Isolated Liver Metastasis: Patients with advanced colorectal cancer with isolated liver metastasis. Primary cancer must be resectable (if no archival exists) and patient must be planned for liver resection with at least 3 cycles of chemotherapy prior to liver surgery.

SUMMARY:
This is a prospective study investigating the disease course of patients with colorectal cancer that have had their cancer spread to their liver. The aim of this study is find potential biomarkers for disease recurrence and therapeutic targets for prognostic information.

DETAILED DESCRIPTION:
Colorectal cancer (CRC), the 2nd leading cause of cancer mortality, often has a pattern of targeting the liver during initial metastases. The Comprehensive Genomic Profiling of Colorectal Cancer Patients with Isolated Liver Metastases to Understand Response and Resistance to Cancer Therapy (COMPARISON) study aims to assess the disease course of CRC by collecting primary tumor and metastatic liver specimens following pre-operative chemotherapy. If relapse occurs following surgical resection of the liver, biopsies will also be done for molecular analysis. As a result, these samples can be analyzed for chemotherapy resistance mechanisms and therapeutic targets to determine potential clinical outcomes for this particular subset of CRC patients.

ELIGIBILITY:
Eligibility Criteria:

1. Patients must have histologically confirmed CRC with isolated liver metastasis
2. Patients must be planned for a hepatic metastasectomy
3. Patients must have received at least 3 cycles of chemotherapy (FOLFOX or FOLFIRI with or without Bevacizumab) prior to the planned hepatic metastasectomy
4. Primary tumor must be considered resectable with a plan for this to either occur concurrently with the liver resection or subsequent to this.
5. If primary has already been resected before liver resection, archival tissue must be available for genomic analysis
6. Patients must be 18yrs of age or older
7. Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

1. Patients with un-resectable or borderline resectable isolated liver metastases as judged by the multidisciplinary hepatobiliary tumor board at PM or BCCA after a course of pre-operative chemotherapy will be excluded
2. Patients with evidence of possible metastatic disease at any sites outside the liver are not eligible
3. Patients with any major co-morbidity or co-morbidities that will render liver resection very high risk in investigator's opinion
4. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
5. Patients with a previous history of another primary cancer treated within 5 years of study entry are not eligible except those with basal cell or squamous cell carcinoma of the skin and intraepithelial neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic colorectal cancer, isolated liver metastases, at least 3 rounds of chemotherapy (FOLFOX or FOLFIRI +/- Bevacizumab) prior to planned liver resection
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Utilization rates of characterized genomic and epigenetic features associated with chemotherapy resistance and tumor recurrence in clinical environments | 5 years

SECONDARY OUTCOMES:
Identification of epigenetic profiles of recurring tumor clones through serial DNA characterization on the NGS platform | 5 years
Identification of epigenetic profiles of recurring tumor clones through serial RNA characterization on the NGS platform | 5 years
Identification of DNA methylation profiles of recurring tumor clones through serial methylome analysis via MethylSeq | 5 years
Non-invasive detection of cfDNA methylation profiles by performing ultra-deep targeted NGS on blood samples | 5 years
Non-invasive detection of cfDNA methylation profiles by performing cfMeDIP-seq on blood samples | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre; Kyaw Aung, MD, Principal Investigator — Princess Margaret Cancer Centre; Daniel Renouf, MD, Principal Investigator — British Columbia Cancer Agency
Locations (2):
- Canada (2):
  - Vancouver Regional Cancer Centre, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario